CLINICAL TRIAL: NCT02168907
Title: Phase I Dose-Escalation Study of CPI-613, in Combination With Bendamustine and Rituximab, in Patients With Relapsed or Refractory B-Cell Non-Hodgkin Lymphoma
Brief Title: CPI-613, Bendamustine Hydrochloride, and Rituximab in Treating Patients With Relapsed or Refractory B-Cell Non-Hodgkin Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow Accruals
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00027759; NCI-2014-01280 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 28114 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2014-06-18; First posted 2014-06-20 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: B-cell Adult Acute Lymphoblastic Leukemia; B-cell Chronic Lymphocytic Leukemia; Cutaneous B-cell Non-Hodgkin Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Intraocular Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Hairy Cell Leukemia; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; Testicular Lymphoma; Waldenström Macroglobulinemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Intraocular Lymphoma; Lymphoma, B-Cell, Marginal Zone; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Hairy Cell; Waldenstrom Macroglobulinemia | interventions — devimistat; Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (CPI-613, bendamustine hydrochloride, rituximab) (Experimental): Patients receive 6,8-bis(benzylthio)octanoic acid intravenously IV over 2 hours on days 1-4 (week 1) and days 1 and 4 (weeks 2 and 3). Patients also receive bendamustine hydrochloride IV over 30 minutes on days 4 and 5 and rituximab on day 5 of week 1. Treatment repeats every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: 6,8-bis(benzylthio)octanoic acid; Drug: bendamustine hydrochloride; Biological: rituximab; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: 6,8-bis(benzylthio)octanoic acid — Given IV
  Other Names: alpha-lipoic acid analogue CPI-613; CPI-613
Drug: bendamustine hydrochloride — Given IV
  Other Names: bendamustin hydrochloride; bendamustine; cytostasan hydrochloride; Treanda
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of CPI-613 (6,8-bis[benzylthio]octanoic acid) when given together with bendamustine hydrochloride and rituximab in treating patients with B-cell non-Hodgkin lymphoma that has come back or has not responded to treatment. Drugs used in chemotherapy, such as 6,8-bis(benzylthio)octanoic acid and bendamustine hydrochloride, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Monoclonal antibodies, such as rituximab, may find cancer cells and help kill them. Giving 6,8-bis(benzylthio)octanoic acid with bendamustine hydrochloride and rituximab may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of CPI-613, when used in combination with bendamustine (bendamustine hydrochloride) and rituximab in patients with relapsed or refractory B-cell non-Hodgkin lymphoma (NHL), who have or have not received hematopoietic cell transplant.

SECONDARY OBJECTIVES:

I. To evaluate response rate (RR) and disease control rate (DCR), derived from the modified International Work Group (IWG) criteria.

II. To evaluate overall survival (OS) and progression-free-survival (PFS), and possible correlation between RR and DCR derived from the modified IWG criteria vs. OS and PFS.

III. To evaluate assessment of bone marrow biopsy, and possible correlation between complete response (CR) vs. bone marrow biopsy assessment (e.g., clear of infiltration of leukemic cells accordingly to morphology, and/or negative on leukemic cells according to immunohistochemistry).

IV. To evaluate safety of the CPI-613 + bendamustine + rituximab combination.

OUTLINE: This is a dose-escalation study of 6,8-bis(benzylthio)octanoic acid.

Patients receive 6,8-bis(benzylthio)octanoic acid intravenously (IV) over 2 hours on days 1-4 (week 1) and days 1 and 4 (weeks 2 and 3). Patients also receive bendamustine hydrochloride IV over 30 minutes on days 4 and 5 and rituximab on day 5 of week 1. Treatment repeats every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically and cytologically confirmed B-cell NHL that has relapsed from, or is refractory to, all standard therapies (including autologous transplantation) known to provide clinical benefit, but have not been treated with bendamustine for their lymphoma
* Must have measurable disease (e.g., a tumor mass > 1 cm)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Expected survival > 3 months
* Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must use accepted contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive or double barrier device) during the study, and must have a negative serum or urine pregnancy test within 1 week prior to treatment initiation
* Fertile men must practice effective contraceptive methods during the study, unless documentation of infertility exists
* At least 2 weeks must have elapsed from any prior surgery
* Aspartate aminotransferase (AST/serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT/serum glutamate pyruvate transaminase [SGPT]) =< 3 x upper normal limit (UNL) (=< 5 x UNL if liver metastases present)
* Bilirubin =< 1.5 x UNL
* Serum creatinine =< 1.5 mg/dL or 133 umol/L
* "International normalized ratio" or INR must be =< 1.5
* No evidence of active infection and no serious infection within the past month
* Mentally competent, ability to understand and willingness to sign the informed consent form

Exclusion Criteria:

* Known cerebral metastases, central nervous system (CNS) or epidural tumor
* Having "currently active" second malignancy unrelated to Hodgkin lymphoma (HL) or NHL, unless they have completed anti-cancer therapy, are in complete response and are considered by their physicians to be at less than 30% risk of relapse
* Patients receiving any other standard or investigational treatment for their cancer, or any other investigational agent for any indication, within the past 2 weeks prior to initiation of treatment with study drugs
* Serious medical illness that would potentially increase patients' risk for toxicity
* Any active uncontrolled bleeding, and any patients with a bleeding diathesis (e.g., active peptic ulcer disease)
* History of abdominal fistula or gastrointestinal perforation =< 6 months prior to treatment with study drugs
* Pregnant women, or women of child-bearing potential not using reliable means of contraception
* Lactating females
* Fertile men unwilling to practice contraceptive methods during the study period
* Any condition or abnormality which may, in the opinion of the investigator, compromise the safety of patients
* Unwilling or unable to follow protocol requirements
* Active heart disease including but not limited to symptomatic congestive heart failure, symptomatic coronary artery disease, symptomatic angina pectoris, symptomatic myocardial infarction or symptomatic congestive heart failure
* Patients with a history of myocardial infarction that is < 3 months prior to registration
* Evidence of active infection, or serious infection within the past month
* Patients with known human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C
* Patients who have received cancer immunotherapy of any type within the past 2 weeks prior to initiation of CPI-613 treatment
* Requirement for immediate palliative treatment of any kind including surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-12; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
MTD of 6,8-bis(benzylthio)octanoic acid, when used in combination with bendamustine hydrochloride and rituximab determined by dose-limiting toxicities graded by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) | 4 weeks
  Will be accomplished by monitoring toxicities and using the dose escalation plan.

SECONDARY OUTCOMES:
Response rate assessed by the modified IWG criteria | Up to 2 years
  The response rate and its 95% confidence interval will be assessed.
Disease control rate assessed by the modified IWG criteria | Up to 2 years
  The DCR and its 95% confidence interval will be assessed.
Overall survival assessed by the modified IWG criteria | Up to 2 years
  OS curves will be plotted using Kaplan-Meier methods.
Progression free survival assessed by the modified IWG criteria | Up to 2 years
  PFS curves will be plotted using Kaplan-Meier methods and median PFS will be examined.
Bone marrow biopsy analysis | Baseline
  Evaluation of bone marrow and possible correlation between CR vs. bone marrow biopsy assessments such as clear of infiltration of leukemic cells accordingly to morphology, and/or negative on leukemic cells according to immunohistochemistry. Correlations will be estimated to examine the relationship between results from bone marrow biopsies and response and time to event results.
Incidence of toxicities graded according to NCI CTCAE | Up to 6 courses
  Will be examined by looking at each toxicity identified earlier in the protocol by grade.

CONTACTS AND LOCATIONS:
Overall Officials: Zanetta Lamar, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States